CLINICAL TRIAL: NCT02886715
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.1% to TAZORAC® (Tazarotene) Cream 0.1% and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing Tazarotene Cream 0.1% to TAZORAC® (Tazarotene) Cream 0.1% and Both to a Placebo Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0454-01-01; 0454 (Other: Fougera Pharmaceuticals Inc.)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)
  Interventions: Drug: Tazarotene Cream 0.1%
- Reference (Active Comparator): TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)
  Interventions: Drug: Tazorac®
- Placebo (Placebo Comparator): Placebo (Vehicle of test product) (Fougera Pharmaceuticals Inc.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tazarotene Cream 0.1% — Tazarotene Cream 0.1% applied to cover the affected areas of the face once daily for 84 +/- 4 days.
  Other Names: Tazarotene
  Arms: Test
Drug: Tazorac® — Tazorac® applied to cover the affected areas of the face once daily for 84 +/- 4 days.
  Other Names: Tazarotene
  Arms: Reference
Drug: Placebo — Placebo (vehicle of the test product) applied to cover the affected areas of the face once daily for 84 +/- 4 days.
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.1% to TAZORAC® (Tazarotene) Cream 0.1% and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Must have a minimum of ≥ 25 non-inflammatory lesions and ≥ 20 inflammatory lesions and ≤ 2 nodulocystic lesions at baseline on the face.
* Must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Have a history of hypersensitivity or allergy to tazarotene, retinoids and/or any of the study medication ingredients.
* Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1110 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela C. Kaplan, Study Director — Fougera Pharmaceuticals Inc.
Locations (23):
- United States (23):
  - Fougera Investigational Site, Tucson, Arizona
  - Fougera Investigational Site, Conway, Arkansas
  - Fougera Investigational Site, Hot Springs, Arkansas
  - Fougera Investigational Site, Anaheim, California
  - Fougera Investigational Site, La Mesa, California
  - Fougera Investigational Site, Long Beach, California
  - Fougera Investigational Site, Los Angeles, California
  - Fougera Investigational Site, North Hollywood, California
  - Fougera Investigational Site, San Diego, California
  - Fougera Investigational Site, San Ramon, California
  - Fougera Investigational Site, Upland, California
  - Fougera Investigational Site, West Covina, California
  - Fougera Investigational Site, Coral Gables, Florida
  - Fougera Investigational Site, Miami, Florida
  - Fougera Investigational Site, Miami Gardens, Florida
  - Fougera Investigational Site, Miramar, Florida
  - Fougera Investigational Site, Sweetwater, Florida
  - Fougera Investigational Site, Plainfield, Indiana
  - Fougera Investigational Site, High Point, North Carolina
  - Fougera Investigational Site, Hazleton, Pennsylvania
  - Fougera Investigational Site, Upper Saint Clair, Pennsylvania
  - Fougera Investigational Site, Chattanooga, Tennessee
  - Fougera Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At Baseline Visit eligible subjects were randomized to the Test, Reference or Placebo product in a 2:2:1 ratio using an interactive response technology (IRT) system
Pre-assignment Details: 1154 subjects were screened for study participation, 1110 subjects were randomized and included in the statistical analyses.
  25 investigative sites randomized subjects into the study.
Period: Overall Study
Arm/Group | Test | Reference | Placebo
Started (Randomized - Safety Population) | 442 | 445 | 223
Modified ITT (mITT) | 421 | 418 | 217
Per Protocol (PP) Population | 346 | 351 | 176
Completed | 378 | 390 | 203
Not Completed | 64 | 55 | 20
Not completed — Non-Compliance With Study Drug | 0 | 2 | 0
Not completed — Adverse Event | 4 | 2 | 0
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Lost to Follow-up | 29 | 26 | 10
Not completed — Pregnancy | 1 | 1 | 1
Not completed — Protocol Violation | 3 | 2 | 1
Not completed — Withdrawal by Subject | 20 | 18 | 5
Not completed — missing | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Placebo | Total
Number analyzed (Participants) | 442 | 445 | 223 | 1110
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Started (Safety Population)
  Years | 22.5 (7.0) | 22.7 (7.0) | 22.5 (7.0) | 22.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Started (Safety Population)
  Participants
    Female | 236 | 215 | 96 | 547
    Male | 206 | 230 | 127 | 563
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Started (Safety Population)
  Participants
    Hispanic or Latino | 265 | 252 | 130 | 647
    Not Hispanic or Latino | 177 | 193 | 93 | 463

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Lesion Counts
Description: Percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts
Time Frame: Week 12
Population: mITT for superiority versus placebo, PP for equivalence versus Reference
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 421 | 418 | 217
percent change | -58.44 (1.33) | -60.07 (1.32) | -53.28 (1.81)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% Confidence Interval for the least-squares mean Test/Reference ratios to be within 80-125%; ANOVA — p-value was no calculated; with treatment and site as fixed effects in the model; Test-to-Reference Ratio = 98.75, 90% CI 2-sided [94.39 to 103.31]
Statistical Analysis 2: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0185, ANOVA; with treatment and site as fixed effects in the model; Mean Difference (Final Values) = -5.17, 95% CI 2-sided [-9.46 to -0.87]

2. Secondary Outcome: Clinical Response of Success
Description: The proportion of subjects with a clinical response of success at week 12, success defined as an Investigator's Global Assessment score that is at least two grades less than the baseline assessment
Time Frame: Week 12
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 421 | 418 | 217
percentage of participants | 20.0 | 23.7 | 15.2

3. Primary Outcome: Change in Non-inflammatory Lesion Counts
Description: Percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts
Time Frame: Week 12
Population: mITT for superiority versus placebo, PP for equivalence versus Reference
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 421 | 418 | 217
percent change | -50.11 (1.27) | -51.99 (1.26) | -45.72 (1.73)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% Confidence Interval for the least-squares mean Test/Reference ratios to be within 80-125%; ANOVA — p-value was no calculated; with treatment and site as fixed effects in the model; Test-to-Reference Ratio = 98.39, 90% CI 2-sided [93.42 to 103.61]
Statistical Analysis 2: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0354, ANOVA; with treatment and site as fixed effects in the model; Mean Difference (Final Values) = -4.39, 95% CI 2-sided [-8.48 to -0.30]

ADVERSE EVENTS:
Time Frame: From baseline to week 12 (end of study)
Arm/Group | Test | Reference | Placebo
All-Cause Mortality (participants affected / at risk) | 0/442 | 0/445 | 0/223
Serious Adverse Events (participants affected / at risk) | 1/442 | 0/445 | 0/223
Other Adverse Events (participants affected / at risk) | 45/442 | 57/445 | 12/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=442) | Reference (N=445) | Placebo (N=223)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=442) | Reference (N=445) | Placebo (N=223)
Application site dryness (General disorders) | 11 | 15 | 2
Application site exfoliation (General disorders) | 7 | 8 | 1
Application site pain (General disorders) | 16 | 9 | 1
Application site pruritus (General disorders) | 5 | 10 | 4
Nasopharyngitis (Infections and infestations) | 5 | 10 | 2
Headache (Nervous system disorders) | 7 | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Fougera' agreements with its investigators may vary. However, Fougera does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT02886715/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT02886715/SAP_001.pdf